CLINICAL TRIAL: NCT07115758
Title: The Impact of Vestibular Versus Trapezoidal Flap Design on Immediate Implants : a Randomized Clinical Trial
Brief Title: Vestibular Versus Trapezoid Flap in Immediate Implants
Acronym: VST
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 24-093
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Immediate Dental Implant Placement; Defect in Alveolar Ridge

STUDY DESIGN:
Intervention Model Description: To address the labial plate of bone defect, a conventional mucoperiosteal flap will be utilized along with guided bone regeneration (GBR). GBR is a surgical technique that involves the use of bone grafts and barrier membranes to reconstruct buccal osseous defects around dental implants
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VST (Experimental): Elaskary Vestibular socket therapy instruments will be used for the intervention, A 1 cm long vestibular access incision at the allocated hopeless tooth will be made at the base of the hopeless tooth to the adjacent teeth. The vestibular pouch will then be dissected in an incisal direction exposing the total socket area and allowing direct access to the socket environment. An immediate implant will be installed using a surgical guide. A membrane shield 1 mm thick will be, trimmed, and tucked through the vestibular access incision starting at 1 mm beyond the socket orifice and reaching to the apical area of the socket. The gap and/ or the defect between the implant body and the shield will then be filled with the same grafting components so the control group. Finally, the vestibular incision will be secured with sutures. The socket will be sealed with a customized healing abutment.
  Interventions: Procedure: control GBR; Procedure: VST
- GBR (Active Comparator): will have a full thickness papilla preservation FLAP, followed by an immediate implant placement using a surgical guide. Then a guided bone regeneration will be achieved by bone graft (autogenous bone chips and xenograft particles and a membrane barrier 1 mm thickness will be applied. The membrane shield then will be stabilized to the apical bone using 2 membrane tacks, customized healing abutment will be connected , then, the elevated flap will be sutured to its original position.
  Interventions: Procedure: control GBR; Procedure: VST

INTERVENTIONS:
Procedure: control GBR — will have a full thickness papilla preservation FLAP, followed by an immediate implant placement using a surgical guide. Then a guided bone regeneration will be achieved by bone graft (autogenous bone chips and xenograft particles and a membrane barrier 1 mm thickness will be applied. The membrane shield then will be stabilized to the apical bone using 2 membrane tacks, customized healing abutment will be connected , then, the elevated flap will be sutured to its original position.
Procedure: VST — Pre extraction procedure:
  Prior to tooth extraction, cone beam computed tomography (CBCT) images will be taken to inspect the overall socket condition.
  All patients will be scanned pre-operatively using an intra-oral scanner (IOS).
  Extraction protocol:
  incisal extraction technique, where atraumatic tooth extraction to the hopeless tooth will be performed using periotomes followed by conventional forceps.

SUMMARY:
The vestibular socket therapy was introduced by Elaskary et al that allowed immediate implant placement and total socket rehabilitation at the same time in class 2 compromised sockets , that showed supreme esthetic and functional predictability over 1,2,3 years of follow up, and showed minimal or no post restorative mid facial recession . The Vestibular socket therapy (VST) entails socket augmentation through a minimally invasive vestibular access incision to allow the delivery of the grafting components thus bypass the deleterious effect of the classic mucoperiosteal flap reflection as well as the deleterious effect of the delay approach, regardless of the degree of socket compromise [6-8].

DETAILED DESCRIPTION:
The concept of promptly replacing teeth using dental implants was introduced many years ago as a way to reduce the time between tooth extraction and the completion of prosthetic restoration. However, immediate implant placement was not recommended by many authors such as Buser D, and Yong , due to the lack of buccal bone, presence of infection, and the continuing post extraction bone remodeling that occurs along both buccal and lingual plates walls of the socket.It has been proposed that the subsequent resorption of the socket walls after tooth extraction should be taken into account when developing any future treatment plan. Furthermore, the labial plate of bone is already compromised in type II extraction socket and is indicated for guided bone regeneration (GBR) such as early placement protocol, using the contour augmentation procedure. Many authors have conducted immediate implant placement using the conventional immediate implant placement via reflecting a mucoperiosteal flap that enabled the accurate socket debridement , total visibility of the socket environment and the ability to graft the buccal osseous defect.To address the labial plate of bone defect, a conventional mucoperiosteal flap will be utilized along with guided bone regeneration (GBR). GBR is a surgical technique that involves the use of bone grafts and barrier membranes to reconstruct buccal osseous defects around dental implants [10]. Typically, this procedure is performed on defects that are equal to or greater than 2 mm in size, such as dehiscence or fenestration defects. Tension-free primary closure will then achieved either on a cover screw or a healing abutment, several flap designs were proposed to minimize the deleterious effect of the classic approach such as papilla preservative incision and buccal esthetic flaps technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients having a hopeless maxillary tooth in the esthetic region missing coronal tooth structure, type II socket (deficient labial plate of bone and intact overlying soft tissues), adequate palatal bone, ≥ 3 mm apical bone to engage the immediately placed implants, thereby achieving optimum primary stability (a minimum of 30 Ncm insertion torque) following tooth extraction.

Exclusion Criteria:

* Smokers, pregnant women, patients with systemic diseases, and history of chemotherapy or radiotherapy within the past 2 years.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Changes in mid facial recession | 6 months after final restoration
  soft tissue stability measured in mm as difference In mid facial recession between pre operative and six months post operative

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - The British university in Egypt, Cairo, New Cairo
  - Faculty of oral and dental medicine the british university in egypt elsherouk, Cairo

IPD SHARING:
Plan to Share IPD: No
study data available upon resonable request due to privacy